CLINICAL TRIAL: NCT02959996
Title: Liposomal Bupivacaine at Cesarean Delivery to Decrease Post-operative Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Malavika Prabhu, Clinical Fellow, Division of Maternal Fetal Medicine, Department of Obstetrics & Gynecology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P002307/MGH
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline will be infiltrated
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Liposomal bupivacaine will be infiltrated
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — liposomal bupivacaine injection in the Pfannenstiel incision
  Other Names: Exparel
  Arms: Intervention
Drug: Placebo — placebo injection in the Pfannenstiel incision
  Arms: Placebo

SUMMARY:
This is a randomized controlled trial to test whether the use of liposomal bupivacaine at the time of cesarean delivery may decrease post-operative pain scores.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. A total of 80 patients will be randomized 1:1 to intervention (liposomal bupivacaine) versus control (placebo solution).

The planned intervention is the infiltration of liposomal bupivacaine (or control) at the time of fascial closure at a Pfannenstiel incision, after the delivery of the infant and repair of the hysterotomy. The procedure to instill the drug is as follows: Once the patient is in the operating room, neuraxial anesthesia will be administered per routine practice. A Pfannenstiel skin incision will be made. The usual cesarean delivery procedure will be performed at the discretion of the surgeon. Once the surgical team is about to begin fascial closure, the study drug will then be infiltrated by a member of the study team, with 50% of the study solution in subcutaneous space and 50% in the fascial plane, taking care to evenly spread the drug in the superior and inferior aspects of the incision. For the fascial infiltration, liposomal bupivacaine will be preferentially infiltrated laterally. The remainder of the cesarean delivery will proceed according to the usual fashion. At any point in the cesarean delivery, the surgeon may chose to administer or withhold ketorolac.

Post-operative pain management will be: intrathecal morphine, scheduled ketorolac 30mg IV x 24h followed by ibuprofen 600mg q6h x 24h, scheduled Tylenol 650mg q6h x 48h, and prn oxycodone 5-10mg q4h. This is the current pain management protocol for postoperative women after cesarean delivery. If Tylenol or NSAIDs are contraindicated, either due to the discretion of the clinical team or pre-existing patient contraindication, these will not be administered but are not a reason for study exclusion.

The investigators plan to enroll 80 patients into this pilot study, 40 per group. This sample size is based on prior data among women who had a cesarean delivery at this institution, and were asked to report their pain scores with activity at 48- and 72- hours after operation. With this sample size, the investigators have 80% power to detect a 1.5 point difference in pain at 48 hours, and 90% power to detect a 1.5 point difference in pain at 72 hours, and account for any protocol violations or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled cesarean delivery via Pfannenstiel incision;
2. Planned neuraxial anesthetic with intrathecal morphine and fentanyl administration.

Exclusion Criteria:

1. Current or prior use of methadone, buprenorphine, or other opioids before cesarean delivery;
2. Contraindication to neuraxial anesthetic;
3. Allergy to local anesthetic;
4. Planned general anesthetic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Barth, Jr, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prabhu M, Clapp MA, McQuaid-Hanson E, Ona S, O'Donnell T, James K, Bateman BT, Wylie BJ, Barth WH Jr. Liposomal Bupivacaine Block at the Time of Cesarean Delivery to Decrease Postoperative Pain: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):70-78. doi: 10.1097/AOG.0000000000002649. PMID 29889750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 patients enrolled in both groups, however 1 patient in the liposomal bupivacaine group was excluded after randomization.
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (3.7) | 35.6 (4.2) | 35.2 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 31 | 33 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
BMI, pre-pregnancy, kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 27.6 (6.4) | 26.2 (5.3) | 26.9 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score With Activity
Description: Pain score with activity. PAIN OUT scale, which is a 0-10 scale, where 10 is more pain.
  2 patients in the liposomal bupivacaine group were discharged prior to 48 hour assessment, therefore denominator for this outcome is 37, not 39
Time Frame: at 48-hours post-operatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 37
units on a scale | 3.5 [2 to 5.5] | 4 [2 to 5]
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Score With Activity
Description: Pain score with activity. PAIN OUT scale, which is a 0-10 scale, where 10 is more pain.
  4 patients in the placebo group and 7 patients in the liposomal bupivacaine group were discharged prior to the 72 hour assessment
Time Frame: at 72 -hours post-operatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 36 | 32
units on a scale | 3 [3 to 6] | 2.5 [2 to 4]
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority; p = .14, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Opioid Use (in Morphine Equivalents)
Description: Total opioid use (in morphine equivalents)
Time Frame: 72-hours post-operatively
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents (MME)
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 39
morphine milligram equivalents (MME) | 78.8 [33.8 to 123.8] | 75 [7.5 to 105]
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Satisfaction With Post-operative Pain Control
Description: PAIN OUT Tool, 0-10 scale, where 0 is not satisfied and 10 is satisfied
Time Frame: 48-hours post-operatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 37
units on a scale | 9 [7 to 10] | 9 [8 to 10]

5. Secondary Outcome: Postoperative Hospital Length of Stay
Description: Postoperative hospital length of stay
Time Frame: 0 to 96 hours postoperatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 39
days | 3.5 (0.5) | 3.4 (1.0)

6. Secondary Outcome: Number of Patients With Wound Complication - Separation, Dehiscence, Infection
Description: Wound complication - separation, dehiscence, infection
Time Frame: 14 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 39
Participants | 3 | 1

7. Secondary Outcome: Number of Patients With Allergic Reaction Attributable to Local Anesthestic
Description: incisional rash, hives, anaphylaxis
Time Frame: 0-96 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 39
Participants | 0 | 0

8. Secondary Outcome: Operative Time of Cesarean Delivery
Description: Operative time of cesarean delivery
Time Frame: Intraoperative time measurement, from skin incision to skin closure. Measured within 24h of admission.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 40 | 39
hours | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.5]

9. Secondary Outcome: Patient Satisfaction With Pain Management at 6w Postpartum
Description: Phone follow up to ascertain satisfaction with pain control, Likert 5 point scale used
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 37 | 36
Participants | 35 | 33

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Placebo | Intervention
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT02959996/Prot_SAP_000.pdf